## Individually Tailored Lighting System to Improve Sleep in Older Adults NCT01855126

November 5, 2018

## **Study Protocol**

The study will be a randomized trial in 50 community-dwelling older adults with early awakening insomnia who live at home, using a within-subject crossover design. The control condition will be a red light mask; the intervention will be a blue light mask (individualized to the patient's light exposure and circadian rhythm). Subjects will use each condition for eight weeks, with the intervention order counterbalanced across subjects, a two-week baseline observation period, and a two-week washout period between the two study conditions.

Outcomes will be assessed at baseline and 8 weeks for all measures except for (a) side effects, adverse effects, and protocol deviations, which will be monitored weekly, and (b) clinical eye examinations, which will be conducted at baseline and at the end of each study condition.